CLINICAL TRIAL: NCT03384004
Title: Effect of Apical Negative Pressure Irrigation System at Cleaning Lateral Canals and Reduction of Periapical Lesions After Endodontic Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KaVo Kerr (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KK-002
Record Dates: First submitted 2017-12-14; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Root Canal Infection
Keywords: Root Canal Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Irrigation Technique 1 (Experimental): Patients randomized into this group will be treated using EndoVac Pure followed by Ultrasonic Irrigation.
  Interventions: Device: Irrigation Technique 1
- Irrigation Technique 2 (Experimental): Patients randomized into this group will be treated using EndoVac Pure only.
  Interventions: Device: Irrigation Technique 2

INTERVENTIONS:
Device: Irrigation Technique 1 — Irrigation of root canals for this group will be performed using EndoVac Pure, an Apical Negative Pressure Endodontic Irrigation System intended for the delivery and evacuation of endodontic irrigation solutions during root canal procedures. The Endovac Pure is a negative pressure system that utilizes negative pressure irrigation so irrigants are suctioned apically from the pulp chamber to the apical terminus and then through the dental office High Volume Evacuation (HVE) valve (Hi-VAC) system. Endovac Pure is designed to be used with Sodium Hypochlorite (NaOCl or bleach) and EDTA (Ethylenediaminetetraacetic acid). This will be followed by Ultrasonic activation of the sodium hypochlorite solution using Minendo II ultrasonic unit.
  Arms: Irrigation Technique 1
Device: Irrigation Technique 2 — Irrigation of root canals for this group will be performed using the EndoVac pure system without Ultrasonic irrigation. The Endovac Pure is a negative pressure system that utilizes negative pressure irrigation so irrigants are suctioned apically from the pulp chamber to the apical terminus and then through the dental office High Volume Evacuation (HVE) valve (Hi-VAC) system. Endovac Pure is designed to be used with Sodium Hypochlorite (NaOCl or bleach) and EDTA (Ethylenediaminetetraacetic acid).
  Arms: Irrigation Technique 2

SUMMARY:
The aim of the present study is to assess with PA x-rays and CBCT scans the volumetric changes in periapical radiolucencies in endodontically treated teeth 1 year after endodontic treatment and evaluate how well the lateral canals are filled after irrigation with the new generation of negative irrigation pressure unit with and without the ultrasonic irrigation.

DETAILED DESCRIPTION:
This is a single center, prospective clinical study conducted in patients who present for routine endodontic therapy. The study has been reviewed and approved by the Institutional Review Board (Ethics Committee) Aspire IRB located at Santee, CA. The clinical investigator will treat patients who present with radiographic evidence of periapical pathology and will randomize the subjects to either negative pressure irrigation system treatment (EndoVac Pure) with ultrasonic irrigation or negative pressure irrigation system treatment (Endovac Pure) without ultrasonic irrigation. All other aspects of the treatment (access, instrumentation and obturation will be according to clinicians conventional clinical judgment. Subjects will have a pre-treatment PA x-ray and CBCT scan before treatment, a PA x-ray at six months and a CBCT scan at one year post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged at least 18 years.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health in the opinion of the investigator or medically qualified designee;
* No clinically significant and relevant abnormalities of medical history or oral examination;
* Absence of any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Single or multi rooted-canal teeth diagnosed with pulp necrosis and symptomatic/ asymptomatic apical periodontitis as tested with routine diagnostics.
* Radiographic evidence of periapical lesion.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Pre-existing oral irritations. b) Recent (within 30 days) gingival/oral surgery. c) Any clinically significant or relevant oral abnormality.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Any subject requiring re-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline - Size of the lesion in the lateral canals at 1 year | 1 year after endodontic therapy
  Evaluate the efficacy of EndoVac Pure at cleaning lateral canals as evidenced by post-treatment CBCT scans.
  CBCT images will be analyzed and the size of the lesion will be measured and will be evaluated.
Change from baseline - Length of lateral canal filled at 6 months and 1 year | 6 months and 1 year post treatment
  The study will also evaluate how well the lateral canals are filled after irrigation with the new generation of negative irrigation pressure unit with and without the ultrasonic irrigation The amount of filling material visualized in each lateral canal will be calculated and expressed as a percentage of linear extension (length of the lateral canal that was filled, in relation to its entire length in mm).
Change from baseline - Area of the lateral canal filled at 6 months and 1 year | 6 months and 1 year post treatment
  The study will also measure the area occupied by the filling material inside the lateral canal in relation to its entire area in mm²).

SECONDARY OUTCOMES:
Change from baseline - Periapical radiographic healing | 6 months and 1 year after endodontic therapy
  Compare the outcome of periapical radiographic healing 6 months and 1 year after endodontic treatment
  The Periapical Radiographs will be analyzed and the size of the lesion will be measured in two dimensions: mesio-distal and coronal-apical. The lesion will be evaluated based on the findings below:
  Evaluation of Radiographic Findings:
  1. Normal periapical structures
  2. Small changes in bone structures (PAI ≤2)
  3. Changes in bone structures (PAI ≥3)
  4. Periodontitis with well- defined radiolucent area
  5. Severe periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: Brett Gilbert, DDS, Principal Investigator — King Endodontics, LLC
Locations (1):
- King Endodontics,LLC, Niles, Illinois, United States

IPD SHARING:
Plan to Share IPD: No